CLINICAL TRIAL: NCT01562535
Title: A Randomized Clinical Trial of Pronation Versus Supination Maneuvers for the Reduction of the Pulled Elbow
Brief Title: A Clinical Trial of Pronation Versus Supination Maneuvers for the Reduction of the Pulled Elbow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Carlos Alberto Cuello-Garcia, Director of the Center for Evidence Based Medicine & Knowledge Translation, Instituto Tecnologico y de Estudios Superiores de Monterey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMBE-ITESM-2
Record Dates: First submitted 2012-03-21; First posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Nursemaid Elbow; Pulled Elbow
Keywords: pulled elbow; nursemaid elbow
MeSH Terms: interventions — Pronation; Supination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pronation group (Experimental): In this group, participants will receive the pronation procedure. The technique is described below
  Interventions: Other: Pronation
- Supination group (Active Comparator): Participants in this group will be performed the supination technique. Description below.
  Interventions: Other: Supination

INTERVENTIONS:
Other: Pronation — In this technique the arm is flexed 90 degrees and a gentle pronation is applied to the arm; then the arm is further flexed to 45 degrees until the clinician feels a "click" in the elbow meaning the re-accommodation of the radial head has been accomplished.
  Other Names: Hyper-pronation technique
  Arms: Pronation group
Other: Supination — The affected arm is in a 90 degrees flexion. The clinician will hold the arm by the elbow and then makes a gentle supination of the affected arm and flexion of the elbow until feeling the "click" and the child is able to move the arm without pain.
  Other Names: Supination technique
  Arms: Supination group

SUMMARY:
Nursemaid elbow or pulled elbow is a condition commonly seen in the emergency department. It is the sudden pull of the radial head (a bone in the elbow) in toddlers. Usually occur when a parent tries to pull the child by the arm and a "clic" or "clunk" is felt with immediate pain and unwilling to move the arm. It is not a dangerous condition although it is distressing for kids and their parents/caretakers.

DETAILED DESCRIPTION:
The usual therapy consists of one of two maneuvers: supination maneuver or pronation maneuver. They both are safe to perform but none of them have been statistically superior over the other. More studies are needed to confirm or discard the tendency of the studies to favor the pronation maneuver.

The investigators intend to perform a randomized trial evaluating which of these techniques is better than the other in terms of returning the mobility of the affected arm and decreasing pain.

ELIGIBILITY:
Inclusion Criteria:

* Pulled elbow suspected in any child presenting one of the following:

  1. History of an adult or bigger person that had pulled the child's elbow non-intentionally
  2. Presence of intense pain at the arrival at the emergency department and unwilling to move the arm.

Exclusion Criteria:

* Any suspect of injury that could be intentional (child abuse)
* Any suspicion child of suffering a possible fracture (the mechanism of the injury was not from pulling the child's arm, the arm presents obvious deformity, ecchymoses, edema, etc.)
* The mechanism was from multiple trauma
* Any chronic disease affecting the adequate bone mineralization (vitamin D deficiency, osteogenesis, etc.)

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Successful reduction | 10 to 20 minutes
  ✦ Patient can move his/her arm without pain in the next 20 minutes after the technique is applied: i.e., the mother asks the child to hold an object (toy) and the toddler can hold it without problem.

SECONDARY OUTCOMES:
Pain of the procedure | 1 to 5 min
  The mother will asses after the protocol is completed the perceived pain on her child from the maneuver. This will be assessed in a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Cuello-Garcia, MD, Principal Investigator — Instituto Tecnologico y de Estudios Superiores de Monterey
Locations (1):
- School of Medicine and Health Sciences, Monterrey, Nuevo León, Mexico